CLINICAL TRIAL: NCT00048750
Title: A Phase 3, Randomized,Double-Blind, Comparative Study of Micafungin (FK463) Versus Placebo as Preemptive Prophylactic Antifungal Therapy in Patients in the Intensive Care Unit
Brief Title: Comparative Study of Micafungin (FK463) Versus Placebo as Prophylactic Antifungal Therapy in the ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr Manager Clinical Trials Registry, Astellas Pharma US, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01-0-124
Record Dates: First submitted 2002-11-06; First posted 2002-11-08 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Invasive Fungal Infections
Keywords: Anti-Fungal Therapy; Preemptive Anti-Fungal Therapy; Invasive Fungal Infection; Micafungin; ICU
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Micafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Micafungin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: Mycamine; FK463
  Arms: 1
Drug: Placebo — IV
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy and safety of intravenous micafungin versus placebo as prophylactic therapy for invasive fungal infections in patients in the intensive care unit considered to be at high risk.

ELIGIBILITY:
Inclusion Criteria

* Meets entry criteria for high risk

Exclusion Criteria

* Evidence of active invasive fungal infection
* Received more than one dose of systemic antifungal agent within 72 hours prior to first dose of study drug
* Known to be HIV positive who have CD4 count less than 500 cells/mm3
* Has life-expectancy of less than 72 hours or moribund

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2003-01; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the incidence of a proven or probable invasive fungal infection, catheter tip fungal infection, or deep incisional surgical site infection during the study | Baseline through one week post-treatment

SECONDARY OUTCOMES:
Assessment of the incidence of patients requiring alternative systemic antifungal therapy to treat suspected infection | Baseline through one week post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (42):
- United States (35):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Oakland, California
  - Orange, California
  - Sacramento, California
  - San Francisco, California
  - Santa Barbara, California
  - Stanford, California
  - Denver, Colorado
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Atlanta, Georgia
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Portland, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Newark, New Jersey
  - Rochester, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Seattle, Washington
- Canada (7):
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Regina, Saskatchewan
  - Saskatoon, Saskatchewan